CLINICAL TRIAL: NCT04762888
Title: Early Detection, Accurate Staging, and Biologic Characterization of HCC With Hybrid 68Ga-PSMA-Dual -Contrast PET/MRI and PET/CT Using Cyclotron-Produced 68Ga
Brief Title: 68Ga-PSMA-Dual-Contrast PET/MRI or PET/CT for Early Detection of Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-006433; NCI-2021-01092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); W81XWH-20 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (68Ga-PSMA PET/MRI or PET/CT) (Experimental): Patients receive 68Ga-PSMA IV over 90 minutes. Patients then undergo PET/MRI over 60 minutes or PET/CT over 30 minutes.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 Gozetotide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — PET/MRI or PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well 68Ga-PSMA PET/MRI or PET/CT works in early detection of liver cancer. 68Gallium-PSMA is a radioactive tracer designed to circulate through the body and attach itself to the prostate- specific membrane antigen (PSMA) protein on liver cancer cells. Magnetic resonance imaging (MRI) is a scan that uses magnetic and radio waves to produce detailed structural information of the organs, tissues, and structures within the body. Positron emission tomography (PET) is an imaging test that helps to measure the information about functions of tissues and organs within the body. A PET scan uses a radioactive drug (tracer) to show this activity. Computed tomography (CT) scan uses X-rays to create images of the bones and internal organs within your body. Combining a PET scan with an MRI or CT scan may help make the images easier to interpret. This trial may help determine if 68Ga- PSMA PET/MRI or PET/CT can improve upon the diagnosis and management of liver cancer in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility and diagnostic performance of gallium Ga 68 gozetotide (68Ga PSMA)-dual contrast PET/MRI for detection and staging of hepatocellular carcinoma (HCC), and to compare it with standard-of-care (SOC) imaging.

II. To identify the biologic correlates of biomarkers derived from 68Ga PSMA-dual contrast PET/MRI with histopathology features and PSMA immunostaining of HCC.

OUTLINE:

Patients receive 68Ga-PSMA intravenously (IV) over 90 minutes. Patients then undergo PET/MRI over 60 minutes or PET/CT over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either an imaging diagnosis of Hepatocellular carcinoma (HCC) by Computed Tomography (CT) or Magnetic Resonance Imaging MRI (Liver Imaging Reporting and Data System [LI-RADS] 5) confirmed by a board-certified abdominal radiologist, or with biopsy-proven HCC
* Subjects who may undergo hepatic surgical resection, liver transplant, or hepatic locoregional therapy (LRT) (e.g., ablation, embolization, etc.)
* No prior treatment for index HCC lesion (surgical resection, liver transplant, hepatic locoregional therapy arm). Patients that have been previously treated with HCC, but have new or reoccurring untreated lesions, are included in the study.
* Male or female with age greater than 18 years, with the capacity and willingness to provide written informed consent.

Exclusion Criteria:

* Patients requiring emergent surgery for a ruptured/bleeding HCC
* Bilirubin > 3.0 mg/dL, which is a contraindication for Gadoxetate, the MRI contrast agent (relevant to positron emission tomography [PET]/MRI)
* Patients with glomerular filtration rate (GFR) < 30 ml/min/1.73m^2, on dialysis, or with acute kidney injury
* Pregnant and/or breast-feeding patients. A negative pregnancy test within 48 hours of the PET scan
* Patients with higher than the weight/size limitations of PET/MRI or PET/CT scanner
* Subjects with history of allergic response to Eovist or Gadavist
* Subjects with known history of claustrophobia
* Subjects with GFR < 30 ml/min/1.73m^2, on dialysis, or with acute kidney injury
* Subjects with a history of severe hypersensitivity to Eovist or Gadavist
* Patients with contraindication to MRI (relevant to PET/MRI):

  * Patients who have a heart pacemaker
  * Patients who have a metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their brain
  * Patients who have implanted devices with magnets
  * Patients who have other implanted electronic devices
  * Patients who have deep brain stimulator
  * Patients who have vagal nerve stimulator
  * Patients with cochlear (ear) or auditory implants

PSMA PET/CT will be an alternative in this study for patients who are unable to undergo PET/MRI for any reason but are otherwise eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of 68Ga-PSMA-dual contrast | Up to 6 weeks
  Using surgical histopathology of resected or biopsied lesions and routine imaging surveillance (for lesions that cannot be resected or biopsied) as the gold standard, we will estimate the diagnostic performance (lesion-level sensitivity, specificity measures, and corresponding 95% confidence intervals) of PET/MRI for hepatic lesions and extra-hepatic metastases, and compare it with standard-of-care (SOC) imaging (MRI and CT) to identify the incremental benefit of PET/MRI.
Correlate biomarkers derived from PET/MRI with PSMA immuno-histochemical (IHC) grading | Up to 6 weeks
  PSMA stained sections will be evaluated by light microscopy for PSMA localization and the entire section reviewed to determine percentage area of PSMA immunostaining as follows: 0 = no staining, 1 = < 5% staining, 2= 5 to 30% staining, 3 = 31 to 60% staining, and 4 = 61-100% staining. Grades 0-2 will be grouped as 'low PSMA expression' and grades 3 and 4 will be grouped as 'high PSMA expression'
Correlate biomarkers derived from PET/MRI with PSMA immuno-histochemical (IHC) grading | Up to 6 weeks
  Intensity of PSMA uptake in hepatic lesions on PET will be graded as follows: grade 1: uptake < normal liver; grade 2: uptake = normal liver; grade 3: uptake > normal liver; grade 4: uptake > spleen or kidneys. For correlation with PSMA IHC scoring, grades 1 and 2 on PET/MRI will be grouped as 'low PSMA expression'. Conversely, grades 3 and 4 will be grouped as 'high PSMA expression'.

CONTACTS AND LOCATIONS:
Overall Officials: Ajit H. Goenka, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT04762888/ICF_000.pdf